CLINICAL TRIAL: NCT01841190
Title: PROGNOSTIC EVALUATION OF SEVERE SEPSIS AND SEPTIC SHOCK. PROCALCITONIN VERSUS DELTA SOFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, MD. COORDINATOR. ICU., Hospital Sao Domingos
Other Study IDs: hsd1509
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-03

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Prognosis; Sepsis; Septic shock; Procalcitonin; SOFA
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PROCALCITONIN
- DELTA SOFA

SUMMARY:
The purpose of this study is to compare the tendency of plasma concentration and clearance of procalcitonin in the first 24 and 48 hours of management of patients with severe sepsis and septic shock with another marker of early prognosis represented by 48 hours delta sofa.

DETAILED DESCRIPTION:
This is a cohort prospective observational study that will include adult patients admitted to a multidisciplinary ICU of a tertiary hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ICU
* severe sepsis and septic shock

Exclusion Criteria:

* Children
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe sepsis and septic shock admitted to a multidisciplinary ICU
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
MORTALITY | 28 DAYS

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

REFERENCES:
- [Derived] de Azevedo JR, Torres OJ, Beraldi RA, Ribas CA, Malafaia O. Prognostic evaluation of severe sepsis and septic shock: procalcitonin clearance vs Delta Sequential Organ Failure Assessment. J Crit Care. 2015 Feb;30(1):219.e9-12. doi: 10.1016/j.jcrc.2014.08.018. Epub 2014 Sep 10. PMID 25241933